CLINICAL TRIAL: NCT03340662
Title: A Phase 1, Open-Label, 4-Part Study to Evaluate the Effect of Food, Cytochrome P 450 Inhibition and Induction on the Pharmacokinetics of CC 122 in Healthy Adult Subjects
Brief Title: Study Evaluating the Effects of Food, Cytochrome P450 Inhibition and Induction on the Pharmacokinetics of CC-122
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CC-122-CP-006; U1111-1203-1818 (Registry Identifier: WHO)
Record Dates: First submitted 2017-11-09; First posted 2017-11-13 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; CC-122; Adult; Phase 1; CYTOCHROME P450
MeSH Terms: interventions — 3-(5-amino-2-methyl-4-oxoquinazolin-3(4H)-yl)piperidine-2,6-dione; Itraconazole; Fluvoxamine; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- CC-122 Alone under fasted conditions (Experimental): Single oral dose of 3 mg CC-122 administered alone under fasted conditions
  Interventions: Drug: CC-122
- CC-122 plus Itraconazole (Experimental): Single oral dose of 3 mg CC-122 alone and with multiple doses of itraconazole.
  Interventions: Drug: CC-122; Drug: Itraconazole
- CC-122 plus Fluvoxamine (Experimental): Single oral dose of 3 mg CC-122 alone and with multiple doses of fluvoxamine.
  Interventions: Drug: CC-122; Drug: Fluvoxamine
- CC-122 plus Rifampin (Experimental): Single oral dose of 3 mg CC-122 alone and with multiple doses of rifampin
  Interventions: Drug: CC-122; Drug: Rifampin

INTERVENTIONS:
Drug: CC-122 — CC-122
Drug: Itraconazole — CYP3A Inhibitor
  Arms: CC-122 plus Itraconazole
Drug: Fluvoxamine — CYP1A2 Inhibitor
  Arms: CC-122 plus Fluvoxamine
Drug: Rifampin — CYP3A Inducer
  Arms: CC-122 plus Rifampin

SUMMARY:
This is a phase 1 open-label 4-part study to evaluate the effect of food, cytochrome P450 inhibition and induction on the pharmacokinetics of CC 122 in healthy adult subjects. Approximately 81 subjects will be enrolled. There will be approximately 24 subjects in Part 1 and approximately 19 subjects in Parts 2, 3, and 4, respectively. Subjects may participate in 1 part only.

DETAILED DESCRIPTION:
This study will consist of 4 parts. Each part has two periods. The parts may be conducted in any order. Subjects may participate in 1 part only.

Each subject will participate in a screening phase, a baseline phase in each study period, a treatment phase in each study period and a follow-up telephone call. Subjects will be screened for eligibility. Eligible subjects will return to the study center on Day -1 of Period 1 and will remain at the study center until the last day of Period 2.

Part 1: On Day 1 of Period 1, eligible subjects will be randomized to 1 of 2 sequences. On Day 1 of each study period, each subject will receive 1 of 2 treatments according to the sequence in which he or she is randomized.

In Part 2, subjects will receive a single dose of CC-122 in Period 1 and, following an appropriate washout, multiple doses of itraconazole plus one dose of itraconazole with CC-122 in Period 2.

In Part 3, subjects will receive a single dose of CC-122 in Period 1 and, following an appropriate washout, multiple doses of fluvoxamine plus one dose of fluvoxamine with CC-122 in Period 2.

In Part 4, subjects will receive a single dose of CC-122 in Period 1 and, following an appropriate washout, multiple doses of rifampin plus one dose of rifampin with CC-122 in Period 2.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject must understand and voluntarily sign an Informed Consent Form (ICF) prior to any study-related assessments/procedures being conducted.
2. Subject is ≥ 18 and ≤ 55 years of age at the time of signing the ICF.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Subject is in good health as determined by a physical exam at screening.
5. Subject agrees to abide by the requirements and restrictions outlined in the CC-122 Pregnancy Prevention Plan for Subjects in Clinical Trials.
6. Female subjects NOT of childbearing potential must:

   a. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle-stimulating hormone [FSH] level of > 40 IU/L at screening).
7. Male subjects must:

   a. Practice true abstinence2 (which must be reviewed on a monthly basis, as applicable, and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or female of childbearing potential (FCBP)3 while participating in the study, during dose interruptions, and for at least 90 days after the last dose of Investigational Product (IP), even if he has undergone a successful vasectomy.
8. Subject has body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
9. Subject has clinical laboratory safety test results that are within normal limits or

   - considered not clinically significant by the Investigator. Platelet count, absolute neutrophil count, and absolute lymphocyte count must be above the lower limit of normal at screening.
10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
11. Subject has a normal or clinically acceptable 12-lead ECG at screening. In addition:

    1. If male, subject has a QTcF value ≤ 430 msec at screening.
    2. If female, subject has a QTcF value ≤ 450 msec at screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject has any hypersensitivity, allergy, or other contraindication to the components of the CC-122, itraconazole, fluvoxamine, or rifampin formulations used in this study (see IB and product labels for relevant information).
5. Subject is a female of childbearing potential, pregnant, or breastfeeding.
6. Subject was exposed to an investigational drug (new chemical entity) within 30 days preceding the first dose administration, or five half-lives of that investigational drug, if known (whichever is longer).
7. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 30 days or 5 terminal half-lives (whichever is longer) prior to the first dose administration.
8. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements, and herbal medicines) within 14 days prior to the first dose administration.
9. Subject has used CYP3A and/or CYP1A2 inducers and/or inhibitors (including St. John's wort) within 30 days prior to the first dose administration.
10. Subject has any surgical or medical condition possibly affecting drug absorption, distribution, metabolism and excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable.
11. Subject donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.
12. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs.
13. Subject has a history of alcohol abuse (as defined by the current version of the DSM) within 2 years before the first dose administration, or positive alcohol screen.
14. Subject has a CYP1A2*1 allele or a CYP3A4*22 allele (PARTS 2, 3, AND 4 ONLY).
15. Subject is known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
16. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self-reported).
17. Subject has received immunization with a live or live attenuated vaccine within 2 months prior to administration of the first dose of IP or is planning to receive immunization with a live or live attenuated vaccine for 2 months after administration of the last dose of IP.
18. Subject is part of the clinical staff personnel or a family member of the clinical site staff.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2018-01-27 (Actual); Study Completion 2018-01-27 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic- Cmax | up to approximately 1 month
  Observed maximum plasma concentration
Pharmacokinetic- AUC 0-∞ | up to approximately 1 month
  Area under the plasma concentration-time curve calculated from time zero extrapolated to infinity

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of treatment
  Number of subjects with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Leon Carayannopoulos, MD, Study Director — Celgene Corporation
Locations (1):
- PPD Phase 1 Clinic, Austin, Texas, United States